CLINICAL TRIAL: NCT04353739
Title: Testing a Self-management Intervention in HIV+ Asian Pacific Americans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Apait Health Center (Other)
Responsible Party: Principal Investigator, Weiti Chen, RN, CNM, PhD, FAAN, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB#20-000580
Record Dates: First submitted 2020-04-14; First posted 2020-04-20 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Self-management
Keywords: family-informed self-management; Asian Pacific Americans
MeSH Terms: interventions — Self-Management

STUDY DESIGN:
Intervention Model Description: Intervention Core Modules: Developed upon the results of the prior studies involving familial relations among APA HIV+ populations, the family-informed self-management intervention has been fully manualized, and has eight modules: (1) psycho-education, (2) cognitive-behavioral management skills training, (3) preparation for disclosure, (4) family relations and support management, (5) anxiety and depressive symptom management, (6) brief mindfulness training, (7) symptom reduction, and (8) the Life-Steps program. The intervention will be delivered via four face-to-face, one-on-one counseling sessions to the participants over 4 weeks. Each module will take on 30 minutes for delivery and each session will deliver two modules in sequence. The primary desired outcome is improved quality of life and diminished viral load.
Who Masked: Participant
Masking Description: There are four data collection points: week 1 (before intervention for immediate treatment (IT) group), week 4 (right after intervention for the IT group, but before intervention for delayed treatment (DT) group), week 7 (after intervention for the DT group), and week 10. Therefore, in this data collection schedule, the IT group will have one-baseline (week 1), two-post-intervention evaluation (week 4), and three and four- follow-ups with 3-week intervals (week 7 and week 10), while the DT group will have 2 baselines (week 1 & week 4), 1 post-intervention evaluation (week 7), and 1 follow-up with a 3-week interval (week 10). Assessment consists of surveying at two times and a dried blood spot test at week 1 and 4.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Treatment (IT) (Experimental): This small RCT will contain two arms, with participants randomly assigned to either the immediate treatment group (IT Group) or the delayed treatment group (DT Group).
  Interventions: Behavioral: Self-Management for HIV-positive Asian Pacific Americans
- Delay Treatment (DT) (Active Comparator): This small RCT will contain two arms, with participants randomly assigned to either the immediate treatment group (IT Group) or the delayed treatment group (DT Group).
  Interventions: Behavioral: Self-Management for HIV-positive Asian Pacific Americans

INTERVENTIONS:
Behavioral: Self-Management for HIV-positive Asian Pacific Americans — Developed upon the results of our prior studies involving familial relations among APA HIV+ populations, the family-informed self-management intervention has been fully manualized and has eight modules: (1) psycho-education, (2) cognitive-behavioral management skills training, (3) preparation for disclosure, (4) family relations and support management, (5) anxiety and depressive symptom management, (6) brief mindfulness training, (7) symptom reduction, and (8) the Life-Steps program.

SUMMARY:
HIV infection rates are on a rapid rise within Asian Pacific Americans (APA) communities, with 80% of new infects being men. The purpose of this study is to adapt and evaluate the feasibility of a 4-session, 4-week family-informed self-management intervention protocol to promote health among APA men with HIV (APAMHIV). Family-informed self-management is a promising intervention to assist APAMHIV in securing family support and promoting health, and hence help address HIV epidemics in this understudied population.

DETAILED DESCRIPTION:
HIV infection rates are on a rapid rise within Asian Pacific Americans (APA) communities, 17% annually, with men comprising 80% of new infections in the United States. Optimal self-management is a key to HIV treatment success, because it may alleviate physical and mental symptoms, promote health behaviors, and therefore enhance quality of life and suppress virus replication. Studies suggested that securing assistance from family members in self-management may be effective in addressing these challenges in APA communities. The purpose of this study is to adapt and evaluate the feasibility of a 4-session, 4-week family-informed self-management intervention protocol to promote health among APA men with HIV (APAMHIV). The scientific premise is, regardless of Asian ethnicity, APA communities often share a more collectivist orientation, such that APA prioritizing their responsibilities to their families over their own individual needs. To preserve the harmony in family, HIV disclosure is often indirect. In previous projects, investigators interviewed an ethnically diverse sample of 40 APAMHIV and 20 family members to explore self- and family- management strategies. The hypothesis is that APAMHIV will receive greater levels of family support and health following the family-informed self-management intervention. This study addresses the critical need to optimize self-management skills among APAMHIV that simultaneously address the needs of APAMHIV with support from their families. The long-term goal is to implement a comprehensive, family-informed self-management intervention for APAMHIV. In this project, researchers will conduct a mixed-methods study with two study phases. In Phase 1, researchers will analyze the available qualitative data from the prior projects to revise the conceptualization of family-informed self-management. Based on the revised conceptualization, researchers will adapt an evidence-based self-management intervention using a modified ADAPT-ITT model. In Phase 2, researchers will conduct a pilot waitlist-controlled clinical trial to test the feasibility, acceptability, and preliminary efficacy of the adapted family-informed self-management intervention among 30 APAMHIV without explicitly involving their family members. This small RCT will contain two arms, with participants randomly assigned to either the immediate treatment group (IT Group) or the delayed treatment group (DT Group). Researchers will evaluate feasibility, acceptability, and preliminary effect sizes, and use the data to revise this family-informed self-management intervention protocol. This will provide the basis for future applications for a fully powered Randomized Controlled Trial of the protocol in the future. Aims are to: 1. Follow the ADAPT-ITT model to culturally adapt an evidence-based family-informed self-management intervention 2. Evaluate the feasibility, acceptability, and preliminary efficacy with a randomized waitlist-controlled trial. And, 3. Finalize the study protocols for future project operations by documenting emerging difficulties and solutions throughout this project implementation.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

1. be at least 18 years of age,
2. be self-identifying as APA,
3. be self-identifying as men,
4. be able to give informed consent to the study,
5. are currently taking ART and
6. be physically well enough to attend counseling sessions and follow-up visits.

Exclusion Criteria:

Participants who:

1. have a significant condition such as neurological or cardiovascular diseases that prevents them from fully participating the study, or
2. are unable to communicate in English or a major Asian language.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life after Self-management intervention | Week 10
  To measure eight domains of health. Questions are a sampling of items from each of the eight domains of health from the SF-36. Each indicator variable is weighted for each of the response choices, minus one.
Biomarker | Week 10
  Viral Load (VL). The VL will be obtained from self-report surveys.
Biomarker | Week 10
  CD4- CD4 will be obtained from self-report surveys.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - APAIT, Los Angeles, California
  - Chinese-American Planning Council., Inc., New York, New York

IPD SHARING:
Plan to Share IPD: Undecided
We will make sure CPC and study participants are willing to share their personal data with researchers. Then, we can release the data.